CLINICAL TRIAL: NCT04219267
Title: Effectiveness of Character Strengths-based Intervention in Enhancing Self-esteem, Quality of Life and Alleviating Depression Among Breast Cancer Patients: A Randomized Controlled Study
Brief Title: Effectiveness of Character Strengths-based Intervention Among Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tingting YAN, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019.429
Record Dates: First submitted 2019-12-20; First posted 2020-01-07 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: self-esteem; quality of life; depression
MeSH Terms: conditions — Breast Neoplasms; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Character strengths-based intervention, 3 sessions every week for three weeks. 30 minutes each session.
  Interventions: Behavioral: character strengths-based intervention
- The control group (Placebo Comparator): Early memories for placebo control, 3 sessions every week for three weeks. 30 minutes each session.
  Interventions: Behavioral: early memories

INTERVENTIONS:
Behavioral: character strengths-based intervention — Character strengths-based intervention (CSI) is one kind of positive psychology interventions. It specifically focuses on character strengths, related activities and exercises assisting individuals to reconnect with their characters and promote self-conceptualization.
  The researcher will develop an education module on CSI based on the previous literatures conducted in China and other countries. Before the RCT, this module will be adapted to Chinese participants. During the intervention, participants in the intervention group will be offered the educational module to learn about strengths, comments around the definition of character strengths and examples of specific strengths.
  Other Names: strengths-based intervention
  Arms: The intervention group
Behavioral: early memories — In early memories, participants will be instructed to write down something from their early memories every day. The memories could be the things happened several days or many years before the writing day. The memories could be participant' travel experiences or food for a day. There are no strict restrictions on the timing or content of these early events.
  Arms: The control group

SUMMARY:
The research design is a randomized control trial to evaluate the effectiveness of character strengths-based intervention in enhancing self-esteem, quality of life and alleviating depression in breast cancer patients. The type of intervention is psychological intervention. Participants in the intervention group will receive character strengths-based intervention. Participants in the control group will receive placebo control care.

DETAILED DESCRIPTION:
The character strengths-based intervention may could enhance self-esteem, quality of life and alleviate depression, but the placebo control care did not do so.

Strengths use is indeed associated with elevated levels of life satisfaction and quality of life. It is positively related to self-esteem and leads to greater self-esteem over time. Moreover, strengths use could help decrease depression in the patients, and has beneficial effect on quality of life. There is a model that examined the mechanism of how strengths use related to enhanced self-esteem, happiness and life satisfaction. Individuals who use their strengths and experience greater levels of life satisfaction is mediated by self-esteem and depression.

Preliminary evidence suggested that character strengths-based intervention has positive impact on psychological well-being include improving self-esteem among women with breast cancer in Spain. However, there is a worldwide paucity of rigorous trials that have evaluated the effectiveness of character strengths-based interventions for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed diagnosis of breast cancer;
* aged above 18 years old;
* native Chinese and proficient in oral mandarin communication;
* agree to participate in the study and offer a written informed consent regarding their voluntary;
* are able to comprehend and complete the questionnaires independently.

Exclusion Criteria:

* suffering from other or multiple life-threatening diseases;
* psychosis (for example, delusional disorder, schizophrenia);
* having participated in any type of group or individual psychological intervention in the past half year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline self-esteem at 2 months,The Rosenberg Self-esteem Scale (RSES) | baseline, 1 and 2 months
  The RSES measures the overall sense of being capable and feeling worthwhile and competent. The Chinese version of RSES will be used in this study. The questionnaire consists of 10 items measured on a five-point Likert scale, higher scores indicating higher self-esteem.

SECONDARY OUTCOMES:
Change from baseline quality of life at 2 months, The Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B, version 4) | baseline, 1 and 2 months
  The Chinese version of FACT-B has undergone cultural adaptation and been used among breast cancer patients in China for many years. The scale consists of 37 items, which are clustered into five domains of quality of life: physical, emotional, social / family, functional well-being and additional concerns of breast cancers, scoring from 0 to 4.
Change from baseline depression at 2 months, The Patient Health Questionnaire 9 (PHQ-9) | baseline, 1 and 2 months
  The Patient Health Questionnaire 9 (PHQ-9) will be used to assess the symptoms of depression by reporting the frequency and the degree of emotional distress in the past two weeks.
Change from baseline character strengths at 2 months, The Chinese Virtues Questionnaire (CVQ) | baseline, 1 and 2 months
  The Chinese Virtues Questionnaire (CVQ) will be used to assess the character strengths of participants. It is the Chinese version of Values in Action Inventory of Strengths (VIA-IS). The CVQ has 96 items. Each question uses five-point Likert scale from "very unlike me" to "very much like me". The higher the score of a character strength, the more prominent the strength of the subject. This scale was developed to examine a person's signature strengths, and has been widely used in adults from various countries.

OTHER OUTCOMES:
Participants' satisfaction with care | 1 month
  Participants' satisfaction with care during the study will be assessed on a five-item checklist developed for this study. Questions such as "Overall, how satisfied are you with the care so far?" will be rated on a five-point Likert scale, ranging from 1 "not at all" to 5 "very much". For each item, higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Chan, PhD, Study Director — The Chinese University of Hongkong; Ka Ming Chow, PhD, Study Director — The Chinese University of Hongkong
Locations (2):
- China (2):
  - Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Abri R, Al-Balushi A. Patient satisfaction survey as a tool towards quality improvement. Oman Med J. 2014 Jan;29(1):3-7. doi: 10.5001/omj.2014.02. PMID 24501659
- [Background] Andrewes HE, Walker V, O'Neill B. Exploring the use of positive psychology interventions in brain injury survivors with challenging behaviour. Brain Inj. 2014;28(7):965-71. doi: 10.3109/02699052.2014.888764. Epub 2014 Mar 21. PMID 24826958
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Background] Carlson LE, Angen M, Cullum J, Goodey E, Koopmans J, Lamont L, MacRae JH, Martin M, Pelletier G, Robinson J, Simpson JS, Speca M, Tillotson L, Bultz BD. High levels of untreated distress and fatigue in cancer patients. Br J Cancer. 2004 Jun 14;90(12):2297-304. doi: 10.1038/sj.bjc.6601887. PMID 15162149
- [Background] Carver CS, Smith RG, Antoni MH, Petronis VM, Weiss S, Derhagopian RP. Optimistic personality and psychosocial well-being during treatment predict psychosocial well-being among long-term survivors of breast cancer. Health Psychol. 2005 Sep;24(5):508-16. doi: 10.1037/0278-6133.24.5.508. PMID 16162045
- [Background] Victoria Cerezo M, Ortiz-Tallo M, Cardenal V, De La Torre-Luque A. Positive psychology group intervention for breast cancer patients: a randomised trial. Psychol Rep. 2014 Aug;115(1):44-64. doi: 10.2466/15.20.PR0.115c17z7. PMID 25153949
- [Background] Chen S, Chiu H, Xu B, Ma Y, Jin T, Wu M, Conwell Y. Reliability and validity of the PHQ-9 for screening late-life depression in Chinese primary care. Int J Geriatr Psychiatry. 2010 Nov;25(11):1127-33. doi: 10.1002/gps.2442. PMID 20029795
- [Background] Cheung YB, Goh C, Thumboo J, Khoo KS, Wee J. Variability and sample size requirements of quality-of-life measures: a randomized study of three major questionnaires. J Clin Oncol. 2005 Aug 1;23(22):4936-44. doi: 10.1200/JCO.2005.07.141. PMID 16051946
- [Background] Ell K, Sanchez K, Vourlekis B, Lee PJ, Dwight-Johnson M, Lagomasino I, Muderspach L, Russell C. Depression, correlates of depression, and receipt of depression care among low-income women with breast or gynecologic cancer. J Clin Oncol. 2005 May 1;23(13):3052-60. doi: 10.1200/JCO.2005.08.041. PMID 15860863
- [Background] Curwood SE, DeGeer I, Hymmen P, Lehmann P. Using strength-based approaches to explore pretreatment change in men who abuse their partners. J Interpers Violence. 2011 Sep;26(13):2698-715. doi: 10.1177/0886260510388283. Epub 2010 Dec 13. PMID 21156680
- [Background] den Heijer M, Seynaeve C, Vanheusden K, Duivenvoorden HJ, Vos J, Bartels CC, Menke-Pluymers MB, Tibben A. The contribution of self-esteem and self-concept in psychological distress in women at risk of hereditary breast cancer. Psychooncology. 2011 Nov;20(11):1170-5. doi: 10.1002/pon.1824. Epub 2010 Aug 4. PMID 20690113
- [Background] Dura-Ferrandis E, Mandelblatt JS, Clapp J, Luta G, Faul L, Kimmick G, Cohen HJ, Yung RL, Hurria A. Personality, coping, and social support as predictors of long-term quality-of-life trajectories in older breast cancer survivors: CALGB protocol 369901 (Alliance). Psychooncology. 2017 Nov;26(11):1914-1921. doi: 10.1002/pon.4404. Epub 2017 Mar 9. PMID 28219113
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Fann JR, Thomas-Rich AM, Katon WJ, Cowley D, Pepping M, McGregor BA, Gralow J. Major depression after breast cancer: a review of epidemiology and treatment. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):112-26. doi: 10.1016/j.genhosppsych.2007.10.008. PMID 18291293
- [Background] Galiano-Castillo N, Ariza-Garcia A, Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Arroyo-Morales M. Depressed mood in breast cancer survivors: associations with physical activity, cancer-related fatigue, quality of life, and fitness level. Eur J Oncol Nurs. 2014 Apr;18(2):206-10. doi: 10.1016/j.ejon.2013.10.008. Epub 2013 Nov 5. PMID 24201014
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Ha EH, Cho YK. The Mediating Effects of Self-Esteem and Optimism on the Relationship between Quality of Life and Depressive Symptoms of Breast Cancer Patients. Psychiatry Investig. 2014 Oct;11(4):437-45. doi: 10.4306/pi.2014.11.4.437. Epub 2014 Oct 20. PMID 25395975
- [Background] Hartl K, Engel J, Herschbach P, Reinecker H, Sommer H, Friese K. Personality traits and psychosocial stress: quality of life over 2 years following breast cancer diagnosis and psychological impact factors. Psychooncology. 2010 Feb;19(2):160-9. doi: 10.1002/pon.1536. PMID 19189279
- [Background] Jassim GA, Whitford DL, Hickey A, Carter B. Psychological interventions for women with non-metastatic breast cancer. Cochrane Database Syst Rev. 2015 May 28;(5):CD008729. doi: 10.1002/14651858.CD008729.pub2. PMID 26017383
- [Background] Koch AK, Rabsilber S, Lauche R, Kummel S, Dobos G, Langhorst J, Cramer H. The effects of yoga and self-esteem on menopausal symptoms and quality of life in breast cancer survivors-A secondary analysis of a randomized controlled trial. Maturitas. 2017 Nov;105:95-99. doi: 10.1016/j.maturitas.2017.05.008. Epub 2017 May 13. PMID 28551083
- [Background] Lytle MC, Vaughan MD, Rodriguez EM, Shmerler DL. Working with LGBT Individuals: Incorporating Positive Psychology into Training and Practice. Psychol Sex Orientat Gend Divers. 2014 Oct 1;1(4):335-347. doi: 10.1037/sgd0000064. PMID 25544947
- [Background] Martin CR, Thompson DR, Chan DS. An examination of the psychometric properties of the Rosenberg Self-Esteem Scale (RSES) in Chinese acute coronary syndrome (ACS) patients. Psychol Health Med. 2006 Nov;11(4):507-21. doi: 10.1080/13548500500407367. PMID 17129926
- [Background] Mustafa M, Carson-Stevens A, Gillespie D, Edwards AG. Psychological interventions for women with metastatic breast cancer. Cochrane Database Syst Rev. 2013 Jun 4;2013(6):CD004253. doi: 10.1002/14651858.CD004253.pub4. PMID 23737397
- [Background] Proyer RT, Gander F, Wellenzohn S, Ruch W. Positive psychology interventions in people aged 50-79 years: long-term effects of placebo-controlled online interventions on well-being and depression. Aging Ment Health. 2014;18(8):997-1005. doi: 10.1080/13607863.2014.899978. Epub 2014 Apr 8. PMID 24712501
- [Background] Reich M, Lesur A, Perdrizet-Chevallier C. Depression, quality of life and breast cancer: a review of the literature. Breast Cancer Res Treat. 2008 Jul;110(1):9-17. doi: 10.1007/s10549-007-9706-5. Epub 2007 Aug 3. PMID 17674188
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Taylor SE, Brown JD. Illusion and well-being: a social psychological perspective on mental health. Psychol Bull. 1988 Mar;103(2):193-210. No abstract available. PMID 3283814
- [Background] Wan C, Zhang D, Yang Z, Tu X, Tang W, Feng C, Wang H, Tang X. Validation of the simplified Chinese version of the FACT-B for measuring quality of life for patients with breast cancer. Breast Cancer Res Treat. 2007 Dec;106(3):413-8. doi: 10.1007/s10549-007-9511-1. Epub 2007 Mar 22. PMID 17377841
- [Background] Woodworth RJ, O'Brien-Malone A, Diamond MR, Schuz B. Web-Based Positive Psychology Interventions: A Reexamination of Effectiveness. J Clin Psychol. 2017 Mar;73(3):218-232. doi: 10.1002/jclp.22328. Epub 2016 Jul 5. PMID 27377826
- [Background] Zhu J, Ebert L, Liu X, Chan SW. A mobile application of breast cancer e-support program versus routine Care in the treatment of Chinese women with breast cancer undergoing chemotherapy: study protocol for a randomized controlled trial. BMC Cancer. 2017 Apr 26;17(1):291. doi: 10.1186/s12885-017-3276-7. PMID 28446141
- [Derived] Yan T, Chow KM, Xiao J, Liang W, Nguyen KT, Choi KC, Chan CWH. Character Strengths-Based Intervention for Enhancing Self-esteem and Quality of Life and Alleviating Depression in Female Patients With Breast Cancer: A Randomized Controlled Trial. Cancer Nurs. 2025 Mar 24. doi: 10.1097/NCC.0000000000001486. Online ahead of print. PMID 40126453
- [Derived] Yan T, Chan CWH, Chow KM, Xiao J, Li M. Development of an evidence-based, theory-driven, and culturally appropriate character strengths-based intervention for breast cancer patients, following the Medical Research Council Framework. Support Care Cancer. 2022 Dec 16;31(1):45. doi: 10.1007/s00520-022-07538-w. PMID 36525147
- [Derived] Yan T, Chan CWH, Chow KM, Li M. Experiences and perception of character strengths among patients with breast cancer in China: a qualitative study. BMJ Open. 2022 Oct 28;12(10):e061994. doi: 10.1136/bmjopen-2022-061994. PMID 36307158